CLINICAL TRIAL: NCT03473756
Title: An International, Multicenter, Phase 1b/2 Study of Rogaratinib (BAY1163877) in Combination With Atezolizumab as First-line Treatment in Cisplatin-ineligible Patients With FGFR-positive Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: Phase 1b/2 Study of Rogaratinib (BAY1163877) in Combination With Atezolizumab in Urothelial Carcinoma
Acronym: FORT-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19131; 2017-001483-38 (EudraCT Number)
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma
Keywords: Locally advanced or metastatic urothelial carcinoma; Bladder cancer; Checkpoint inhibition; FGFR inhibition
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Rogaratinib; atezolizumab

STUDY DESIGN:
Masking Description: Part A is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rogaratinib + Atezolizumab in Part A (Experimental): Part A: Part A is conducted in patients who are cisplatin-ineligible and have had no prior systemic treatment for locally advanced or metastatic disease.
  Patients will receive rogaratinib plus atezolizumab combination treatment.
  Interventions: Drug: Rogaratinib (BAY1163877); Drug: Atezolizumab

INTERVENTIONS:
Drug: Rogaratinib (BAY1163877) — Part A:Rogaratinib will be administered orally until disease progression, unacceptable toxicity or consent withdrawal. The starting dose of 800 mg b.i.d. will be confirmed using a dose selection design.
Drug: Atezolizumab — Part A: A fixed dose of 1200 mg atezolizumab will be administered through intravenous (i.v.) infusion on Day 1 of each 21-day cycle until disease progression, unacceptable toxicity or consent withdrawal.

SUMMARY:
FORT-2 is designed to evaluate safety, efficacy, RP2D and PK of rogaratinib in combination with atezolizumab in patients with untreated FGFR-positive urothelial carcinoma. The study originally comprised two separate parts: Phase 1b (Part A) and Phase 2 (Part B). The study parts differ in design, objectives, and treatment.

The primary objectives of this Phase 1b study (Part A) are to determine the safety, tolerability, RP2D and pharmacokinetics of rogaratinib in combination with atezolizumab in these patients.

The primary objective of the Part B is to compare progression-free survival (PFS) according to RECIST v1.1 of rogaratinib in combination with atezolizumab over placebo in combination with atezolizumab in untreated patients with FGFR-positive locally advanced or metastatic urothelial carcinoma.

Of note, patients who participate in Part A are not allowed to participate in Part B.

Part B will be initiated once the data from Part A supports continuation of the study, even if this occurs prior to primary completion of Part A. The sponsor may decide not to continue the study as a whole after completion of Part A if the data do not support further development.

Part B of the study will no longer be conducted.

ELIGIBILITY:
Inclusion criteria:

* Existence of archival or fresh tumor biopsy specimen for FGFR1/3 mRNA expression testing
* High FGFR1 or 3 mRNA expression levels (RNAscope score of 3+ or 4+) in archival or fresh tumor biopsy specimen
* Documented locally advanced (T4, any N; or any T, N2-3) or metastatic urothelial carcinoma (transitional cell carcinoma) including urinary bladder, renal pelvis, ureters, urethra, meeting all of the following criteria:
* No prior systemic treatment for locally advanced or metastatic urothelial carcinoma. For patients who received prior adjuvant/neoadjuvant chemotherapy or chemo-radiation for urothelial carcinoma, a treatment-free interval > 12 months between the last treatment administration and the date of recurrence is required in order to be considered treatment-naïve in the metastatic setting. Prior local intra-vesical chemotherapy or prior local immunotherapy is allowed if completed at least 4 weeks before the first study drug administration. Regionally available standard of care options must be considered for all patients.
* Ineligibility for cisplatin-based chemotherapy as defined by any one of the following criteria:

  * Impaired renal function (GFR > 30 but < 60 mL/min/1.73 m2) according to the modification of diet in renal disease (MDRD) abbreviated formula
  * A Hearing loss (measured by audiometry) of > 25 dB at two contiguous test frequencies in at least one ear.
  * Grade ≥ 2 peripheral neuropathy (i.e. sensory alteration or paresthesia including tingling)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1.

Exclusion criteria:

* Active symptomatic or untreated brain metastases as determined by CT or MRI evaluation during screening and prior radiographic assessment.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, granulomatosis with polyangiitis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* History or current condition of an uncontrolled cardiovascular disease including any of the following conditions:

  * Congestive heart failure (CHF) NYHA Class 2 or greater, unstable angina (symptoms of angina at rest) or
  * New-onset angina (within last 3 months before the first study drug administration)
  * Myocardial infarction (MI) within past 6 months before the first study drug administration
  * Unstable cardiac arrhythmias requiring anti-arrhythmic therapy.
* Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or known left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Current diagnosis of any retinal disorders including retinal detachment, retinal pigment epithelial detachment (RPED), serous retinopathy or retinal vein occlusion.
* Current evidence of endocrine alteration of calcium phosphate homeostasis (e.g. parathyroid disorder, history of parathyroidectomy, tumor lysis, tumoral calcinosis, paraneoplastic hypercalcemia).
* Concomitant therapies that are known to increase serum calcium or phosphate levels (i.e. antacids, phosphate-containing laxatives oral/rectal, potassium phosphate) and that cannot be discontinued or switched to a different medication before the first study drug administration
* Treatment with systemic corticosteroids or other systemic immunosuppressant medications within 2 weeks before the first study drug administration, or anticipated requirement for systemic immunosuppressive medications during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (4):
  - University of Arizona Cancer Center, Tucson, Arizona
  - UChicago Medicine Comprehensive Cancer Center - Hyde Park, Chicago, Illinois
  - Barbara Ann Karmanos Cancer Institute - Detroit Headquarters, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Austria (4):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Krankenhaus der Barmherzigen Brüder, Vienna, Vienna
  - Uniklinikum Salzburg - Landeskrankenhaus, Salzburg
  - Universitätsklinikum AKH Wien, Vienna
- France (3):
  - Institut Bergonie - Unicancer Nouvelle Aquitaine, Bordeaux
  - Centre Oscar Lambret - Lille, Lille
  - Institut de Cancérologie de l'Ouest - Saint Herblain, Saint-Herblain
- Germany (3):
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
- Italy (5):
  - Azienda Ospedaliero Universitaria di Modena, Modena, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Europeo di Oncologia s.r.l - Sviluppo di nuovi farmaci per Terapie Innovative, Milan, Lombardy
  - Istituto Oncologico Veneto, Padua, Veneto
  - A.O.U.I. Verona, Verona, Veneto
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- South Korea (3):
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul
- Spain (4):
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Ramón y Cajal | Oncología, Madrid
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Sweis RF, Gajate P, Morales-Barrera R, Lee JL, Necchi A, de Braud F, Penel N, Grunwald V, Maruzzo M, Meran J, Ishida TC, Bao W, Zhou Y, Ellinghaus P, Rosenberg JE. Rogaratinib Plus Atezolizumab in Cisplatin-Ineligible Patients With FGFR RNA-Overexpressing Urothelial Cancer: The FORT-2 Phase 1b Nonrandomized Clinical Trial. JAMA Oncol. 2024 Nov;10(11):1565-1570. doi: 10.1001/jamaoncol.2024.3900. Epub 2024 Sep 19. PMID 39298147
- [Derived] Grunewald S, Politz O, Bender S, Heroult M, Lustig K, Thuss U, Kneip C, Kopitz C, Zopf D, Collin MP, Boemer U, Ince S, Ellinghaus P, Mumberg D, Hess-Stumpp H, Ziegelbauer K. Rogaratinib: A potent and selective pan-FGFR inhibitor with broad antitumor activity in FGFR-overexpressing preclinical cancer models. Int J Cancer. 2019 Sep 1;145(5):1346-1357. doi: 10.1002/ijc.32224. Epub 2019 Mar 13. PMID 30807645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 30 study centers in 8 countries (4 in Austria, 3 in France, 3 in Germany, 5 in Italy, 4 in Japan, 3 in South Korea, 4 in Spain, and 4 in the US) between 15 May 2018 (first informed consent) and 10 July 2024 (last participant last visit).
  Only Part A of the study was completed. Part B was not started in line with the protocol. The decision not to conduct Part B was not related to safety concerns but was based on an overall strategic business decision
Pre-assignment Details: A total of 54 FGFR mRNA-positive subjects (35.3%) successfully completed the prescreening. Of these, 37 subjects (68.5%) completed the screening and were assigned to treatment and 31.5% prematurely discontinued the screening: 29.6% due to screening failure and 1.9% (1 subject) due to withdrawal by subject.
Groups:
- Rogaratinib 800 mg BID + Atezolizumab: Participants receiving 800 mg Rogaratinib twice daily plus Atezolizumab
- Rogaratinib 600 mg BID + Atezolizumab: Participants receiving 600 mg Rogaratinib twice daily plus Atezolizumab
Period: Overall Study
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
Started | 11 | 26
Completed | 1 | 0
Not Completed | 10 | 26
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Adverse Event | 6 | 7
Not completed — Lack of Efficacy | 3 | 10
Not completed — Physician Decision | 0 | 2
Not completed — End of study treatment | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab | Total
Number analyzed (Participants) | 11 | 26 | 37
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 2 | 2 | 4
  From 65-84 years | 9 | 23 | 32
  85 years and over | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 9 | 23 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 23 | 32
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities(DLTs)
Time Frame: Up to 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
Number analyzed (Participants) | 11 | 26
Participants | 1 | 4

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: up to 90 days after the last study medication intake, an average of 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
Number analyzed (Participants) | 11 | 26
Participants | 11 | 26

3. Primary Outcome: Number of Participants With Drug-related TEAEs
Time Frame: up to 90 days after the last study medication intake, an average of 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
Number analyzed (Participants) | 11 | 26
Participants | 11 | 26

4. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events(TESAEs)
Time Frame: up to 90 days after the last study medication intake, an average of 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
Number analyzed (Participants) | 11 | 26
Participants | 8 | 14

5. Secondary Outcome: Objective Response Rate(ORR)
Description: Objective response rate (ORR) was defined as the percentage of patients with complete response (CR) or partial response (PR). Patients for whom best overall tumor response was not CR or PR, as well as patients without any post-baseline tumor assessment were considered non-responders. For all patients, the best overall tumor response was determined locally by investigators using the RECIST (Response Evaluation Criteria In Solid Tumors) criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
Number analyzed (Participants) | 11 | 26
Participants
  complete response | 1 | 4
  partial response | 1 | 10
  no response | 9 | 12

6. Secondary Outcome: Maximal Plasma Concentration (Cmax) of Rogaratinib
Time Frame: At cycle 1 Day 1
Measure: Geometric Mean (Standard Deviation); unit: µg/l
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
Number analyzed (Participants) | 11 | 25
µg/l | 13207.846 (1.379) [lower limit 1.379] | 10372.864 (1.404) [lower limit 1.404]

7. Secondary Outcome: Area Under the Rogaratinib Concentration Versus Time Curve (AUC)
Time Frame: At cycle 1 Day 1, 0-t(last)
Measure: Geometric Mean (Standard Deviation); unit: µg*h/l
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
Number analyzed (Participants) | 11 | 25
µg*h/l | 59187.389 (1.513) | 45768.289 (1.449)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were defined as any event arising or worsening after the start of study drug administration up to 90 days after the last study medication intake, an average of 60 days
Arm/Group | Rogaratinib 800 mg BID + Atezolizumab | Rogaratinib 600 mg BID + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 9/11 | 11/26
Serious Adverse Events (participants affected / at risk) | 8/11 | 14/26
Other Adverse Events (participants affected / at risk) | 11/11 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rogaratinib 800 mg BID + Atezolizumab (N=11) | Rogaratinib 600 mg BID + Atezolizumab (N=26)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0)
Renal function test abnormal (Investigations) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Renal cyst aspiration (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rogaratinib 800 mg BID + Atezolizumab (N=11) | Rogaratinib 600 mg BID + Atezolizumab (N=26)
Anaemia (Blood and lymphatic system disorders) | 4 (12) | 4 (14)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Keratopathy (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1)
Maculopathy (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 2 (2)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 4 (6)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 2 (2)
Xerophthalmia (Eye disorders) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Corneal toxicity (Eye disorders) | 1 (1) | 0 (0)
Ocular rosacea (Eye disorders) | 0 (0) | 1 (1)
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 (0) | 1 (2)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 1 (2)
Retinoschisis (Eye disorders) | 0 (0) | 1 (1)
Serous retinopathy (Eye disorders) | 0 (0) | 4 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (8)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (20) | 16 (51)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 7 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (5)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral lichen planus (Gastrointestinal disorders) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (7) | 10 (15)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (4)
Anal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue erosion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (13) | 7 (11)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (6) | 7 (7)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (6) | 11 (26)
Chills (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Hyperpyrexia (General disorders) | 0 (0) | 1 (4)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (3) | 2 (4)
Pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 5 (5)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (13) | 7 (10)
Early satiety (General disorders) | 0 (0) | 1 (1)
Secretion discharge (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 2 (2)
Cystitis (Infections and infestations) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (2)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 4 (5)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (8) | 9 (29)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Herpes dermatitis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (3) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Klebsiella urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (13) | 8 (11)
Stoma site ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 3 (7) | 5 (38)
Aspartate aminotransferase increased (Investigations) | 1 (22) | 6 (7)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 3 (14) | 2 (4)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 3 (4)
Weight decreased (Investigations) | 1 (2) | 3 (3)
Blood phosphorus increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (3)
Lipase increased (Investigations) | 1 (1) | 6 (39)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Calcium phosphate product increased (Investigations) | 2 (4) | 0 (0)
Renal function test abnormal (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 1 (2)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST-T segment abnormal (Investigations) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 (5) | 15 (45)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (6) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (7) | 8 (12)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 6 (11)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (8)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 4 (6)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (3)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (7)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (14)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (10) | 5 (8)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (12)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Astringent therapy (Surgical and medical procedures) | 0 (0) | 1 (4)
Erythromelalgia (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (2)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03473756/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT03473756/SAP_001.pdf